CLINICAL TRIAL: NCT01746706
Title: Can the Assessment of the Subhippocampal Region Contribute to the Detection of Early Diagnosis of Alzheimer's Disease?
Brief Title: Can the Assessment of the Subhippocampal Region Contribute to the Detection of Early Diagnosis of Alzheimer's Disease? A Validation Study Using PET With Florbetapir (AV-45).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011 A00383-38
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients (Experimental)
  Interventions: Device: PET amyloid tracer (Florbetapir F18 AV45 F18
- volunteers (Experimental)
  Interventions: Device: PET amyloid tracer (Florbetapir F18 AV45 F18

INTERVENTIONS:
Device: PET amyloid tracer (Florbetapir F18 AV45 F18

SUMMARY:
Reliable diagnosis of Alzheimer's Disease (AD) at the predementia stage is currently considered to be a priority for research, as disease modifying therapies are being evaluated. Many studies focus on the functional and morphological assessment of the hippocampal formation. However, neurofibrillary tangles, associated with cognitive deficits, initially affect the anterior subhippocampal cortex (transentorhinal, entorhinal and perirhinal cortex) before reaching the hippocampus. Studies from our group have tried to investigate if the assessment of subhippocampal regions using cognitive tools and neuroimaging techniques could contribute to the diagnosis of AD at a very early stage.

In a previous project, the investigators included 40 patients with single domain amnestic MCI (Mild Cognitive Impairment), known to be at high risk for AD and demonstrated that aMCI patients with a profile of subhippocampal dysfunction (impaired performance on a visual recognition memory task) display other clinical as well as imaging profiles of patients with early AD using MRI and SPECT. Longitudinal follow-up data in these patients is currently under way. Preliminary data indicates that evaluating the subhippocampal region using visual recognition tasks is highly predictive of AD over 6 years.

The aim of this project is to obtain additional diagnostic data using a PET amyloid tracer (Florbetapir F18 AV45 F18), an in-vivo marker of one of the neuropathological lesions that define AD, of in order to enhance diagnostic accuracy AD in these patients. This approach will validate the hypothesis as to whether the assessment of subhippocampal dysfunction can contribute to the early diagnosis of AD.

ELIGIBILITY:
Inclusion Criteria:

patients:

* - A score in the MMS (Folstein and al ., on 1975, French version subjected to consensus of Greco). 24 for the level subjects I (less than 5 years of study), 26 and more for the others, the autonomy in the everyday life,
* A lower normal IADL < = 1/4 (Lawton and Brody, on 1969, version 4 items),
* A complaint mnemonic of the patient
* A lower performance of 1,5 standard deviation in the standard in the reminder(abseiling) postponed from the sub-test of logical memory(report) of the WMS-III and/or in the free reminder(abseiling) postponed from the test(event) of the California Verbal Learning Test.

volunteers:

* 50-80-year-old and presented an educational level sailed in that of the patients,
* a MMS upper to 24 for the level subjects I (5 years of study), 26 and more for the levels 2 and 3,
* an Autonomy of the everyday life,
* normal IADL = 0/4
* did not present mnemonic complaint,
* a performance normal for the reminder postponed from the subtest of logical memory of the WMS-III and for the free reminder(abseiling) postponed from the test(event) of the California Verbal Learning Test.

Exclusion Criteria:

* Incapacitated to realize the examination by FART because of medical intercurrent affections. There are this day no contraindications in the product Florbetapir used for the TEPscan.
* The persons under protection of justice cannot be included, because the law forbids their participation biomedical researches.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-10; Primary Completion 2015-11 (Actual); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
the assessment of subhippocampal dysfunction | 24month
  PET amyloid tracer (Florbetapir F18 AV45 F18)

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique Hopitaux De Marseille; mira DIDIC, Principal Investigator — AP HM
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France